CLINICAL TRIAL: NCT01216384
Title: A Randomised, Double-blind (Within Dose Groups), Parallel Group, Placebocontrolled Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Rising Doses (50 mg, 200 mg, 400 mg) of BI 671800 HEA in Chinese Healthy Male Volunteers and Multiple Rising Doses (50 mg b.i.d., 200 mg b.i.d., 400 mg b.i.d.) of BI 671800 HEA in Japanese Healthy Male Volunteers
Brief Title: Single Rising Dose (SRD), Multiple Rising Dose (MRD) Study of BI 671800 in Healthy Asian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1268.15
Record Dates: First submitted 2010-10-01; First posted 2010-10-07 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Asthma; Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Asthma; Rhinitis, Allergic, Perennial | interventions — BI 671800

ARMS (2):
- BI 671800 active (Experimental): SRD part: 3 dose groups each consisting of 12 subjects (9 active, 3 placebo), subjects receive single dose. MRD part: 3 dose groups each consisting of 12 subjects (9 active, 3 placebo), subjects receive single dose followed by multiple doses with a PK sampling interval in between.
  Interventions: Drug: BI 671800
- Placebo (Placebo Comparator): 3 subjects will receive placebo in each of the 3 doses in the SRD part and 3 doses in the MRD part
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: BI 671800 — In the SRD part subjects will receive a single dose and in the MRD part subjects will receive a total of 14 doses.
  Arms: BI 671800 active
Drug: placebo — Subjects will receive according to the dose group matching number of placebo tablets
  Arms: Placebo

SUMMARY:
The primary objective of the current study is to investigate the safety and tolerability of BI 671800 HEA in healthy Chinese male volunteers following single oral administration, and healthy Japanese male volunteers following single oral administration and multiple administrations.

ELIGIBILITY:
Inclusion criteria:

1. Healthy
2. Chinese ethnicity for single rising dose (SRD) part, Japanese Ethnicity for multiple rising dose (MRD) part.
3. Age >= 20 and age =< 50
4. Body Mass Index (BMI) >=18.5 and BMI =< 25 kg/m2
5. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion criteria:

1. Any finding of the medical examination (including blood pressure (BP), pulse rate (PR) and electrocardiogram (ECG)) deviating from normal and of clinical relevance according to the investigators medical judgement
2. Any evidence of a clinically relevant concomitant disease
3. Intake of drugs with long half life (>24 hour) within at least one month or less than 10 half-lives of the respective drug prior to administration

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Physical examination | up to 4 days for SRD part and up to 15 days for MRD part
Vital signs; Blood Pressure(BP) | up to 4 days for SRD part and up to 15 days for MRD part
Vital signs; Pulse rate(PR) | up to 4 days for SRD part and up to 15 days for MRD part
12-lead Electrocardiogram (ECG) | up to 4 days for SRD part and up to 15 days for MRD part
Clinical laboratory tests (Hematology) | up to 4 days for SRD part and up to 15 days for MRD part
Clinical laboratory tests (Clinical chemistry) | up to 4 days for SRD part and up to 15 days for MRD part
Clinical laboratory tests (Urinalysis) | up to 4 days for SRD part and up to 15 days for MRD part
Adverse events | up to 4 days for SRD part and up to 15 days for MRD part

SECONDARY OUTCOMES:
SRD Part, Cmax (maximum measured concentration of the analyte in plasma) BI 671800 and BI 600957 | up to 4 days
SRD Part, tmax (time from dosing to maximum measured concentration), BI 671800 and BI 600957 | up to 4 days
SRD Part, AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time point t1 to time point t2), BI 671800 and BI 600957 | up to 4 days
SRD Part, AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable concentration at tz) BI 671800 and BI 600957 | up to 4 days
SRD Part, AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity), BI 671800 and BI 600957 | up to 4 days
SRD Part, %AUCtz-infinity (the percentage of the AUC 0-infinity that is obtained by extrapolation), BI 671800 and BI 600957 | up to 4 days
SRD Part, λz (terminal rate constant in plasma) ), BI 671800 and BI 600957 | up to 4 days
SRD Part, t1/2 (terminal half-life of the analyte in plasma) BI 671800 and BI 600957 | up to 4 days
SRD Part, MRTpo (mean residence time of the analyte in the body after oral administration) BI 671800 and BI 600957 | up to 4 days
SRD Part, CL/F (apparent clearance of the analyte in plasma after oral administration); only BI671800 | up to 4 days
SRD Part, Vz/F (apparent volume of distribution during the terminal phase λ z following an oral dose); only BI 671800 | up to 4 days
MRD Part , Cmax (maximum measured concentration of the analyte in plasma) BI 671800 and BI 600957 | day1 Visit2, day1 Visit3
MRD Part, tmax (time from dosing to maximum measured concentration), BI 671800 and BI 600957 | day1 Visit2, day1 Visit3
MRD Part, AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time point t1 to time point t2), BI 671800 and BI 600957 | day1 Visit2, day1 Visit3
MRD Part, AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable concentration at tz), BI 671800 and BI 600957 | day1 Visit2, day1 Visit3
MRD Part, AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) , BI 671800 and BI 600957 | day1 Visit2, day1 Visit3
MRD Part, %AUCtz-infinity (the percentage of the AUC 0-infinity that is obtained by extrapolation), BI 671800 and BI 600957 | day1 Visit2, day1 Visit3
MRD Part, λz (terminal rate constant in plasma) ), BI 671800 and BI 600957 | day1 Visit2, day1 Visit3
MRD Part, t1/2 (terminal half-life of the analyte in plasma) BI 671800 and BI 600957 | day1 Visit2, day1 Visit3
MRD Part, MRTpo (mean residence time of the analyte in the body after oral administration) BI 671800 and BI 600957 | day1 Visit2, day1 Visit3
MRD Part, CL/F (apparent clearance of the analyte in plasma after oral administration); only BI671800 | day1 Visit2, day1 Visit3
MRD Part, Vz/F (apparent volume of distribution during the terminal phase λz following an oral dose); only BI 671800 | day1 Visit2, day1 Visit 3
MRD Part, Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ, BI 671800 and BI 600957 | up to 12 days
MRD Part, tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) BI 671800 and BI 600957 | up to 12 days
MRD Part, Cmin,ss (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) BI 671800 and BI 600957 | up to 12 days
MRD Part,tmin,ss (time from last dosing to minimum concentration of the analyte in plasma at steady state) BI 671800 and BI 600957 | up to 12 days
MRD Part,Cpre,ss (predose concentration of the analyte in plasma immediately before administration of dose at steady state) BI 671800 and BI 600957 | up to 12 days
MRD Part,AUCt1-t2,ss (area under the concentration-time curve of the analyte in plasma at steady state over the time interval t1 to t2) BI 671800 and BI 600957 | up to 12 days
MRD Part,AUC τ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) BI 671800 and BI 600957 | up to 12 days
MRD Part,λz ,ss (terminal rate constant in plasma at steady state) BI 671800 and BI 600957 | up to 12 days
MRD Part,t1/2,ss (terminal half-life of the analyte in plasma at steady state) BI 671800 and BI 600957 | up to 12 days
MRTpo,ss (mean residence time of the analyte in the body at steady state after xx administration) BI 671800 and BI 600957 | up to 12 days
CL/F,ss (apparent clearance of the analyte in the plasma at steady state following extravascular multiple dose administration); only BI 671800 | up to 12 days
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration); only BI 671800 | up to 12 days
Accumulation ratios RA,Cmax, 13 based on Cmax after the first dose and at steady state | up to 12 days
Accumulation ratios RA,AUC,13 based on AUC τ after the first dose and at steady state | up to 12 days
Linearity index (LI) of the analyte in plasma | up to 12 days
AUEC0-24,N absolute inhibition of eosinophil shape change: area under the absolute inhibition of shape change-time curve after the Nth dose of BI 671800 HEA | up to day 9
AUEC0-24,N percent inhibition of eosinophil shape change: area under the percent inhibition of shape change - time curve after the Nth dose of BI 671800 | up to day 9

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1268.15.8201 Boehringer Ingelheim Investigational Site, Seoul, South Korea